CLINICAL TRIAL: NCT01656720
Title: A Multi-centre, Phase II, Double-blind, Randomised, Placebo-controlled, Parallel Group, Dose-ranging Study in Patients With Faecal Incontinence; to Evaluate the Efficacy, Safety and Tolerability of Locally Applied NRL001 Over an 8 Week Treatment Period
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRL001-01/2011 (SEFI)
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Faecal Incontinence
Keywords: Faecal Incontinence; Suppository; Wexner score
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Placebo 2g Suppository
  Interventions: Drug: Placebo
- NRL001 5mg (Active Comparator): 5mg NRL001 in a 2g suppository
  Interventions: Drug: 1R, 2S-methoxamine hydrochloride
- NRL001 7.5mg (Active Comparator): 7.5mg NRL001 in a 2g suppository
  Interventions: Drug: 1R, 2S-methoxamine hydrochloride
- NRL001 10mg (Active Comparator): 10mg NRL001 in a 2g suppository
  Interventions: Drug: 1R, 2S-methoxamine hydrochloride

INTERVENTIONS:
Drug: 1R, 2S-methoxamine hydrochloride
  Other Names: NRL001
  Arms: NRL001 10mg; NRL001 5mg; NRL001 7.5mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of NRL001 in the treatment of faecal incontinence, compared against placebo

ELIGIBILITY:
Inclusion Criteria:

* An ultrasound assessment of the internal anal sphincter within the previous 12 months confirming an intact circular internal sphincter with minimal scars (maximum 60 degrees scarring circumferentially).
* Diagnosis of faecal incontinence with a Wexner score of 8 - 20 inclusive at Visit 1 - Screening Visit.
* Historical clinical evidence (past 6 months prior to Visit 1 - Screening Visit) of faecal incontinence episodes (solids, liquid, gas or mucus).
* Greater than or equal to two faecal incontinence episodes (solids, liquid, gas or mucus) per week during the 4 week historical period prior to Visit 1 - Screening Visit.
* Able and willing to receive rectal examinations and treatments.
* Patients must be aged >18 without significant acute or uncontrolled chronic disease.
* Patients must understand the purpose and risks of the study and be able to provide written informed consent and willing, able and competent to complete the entire study and comply with study instructions as defined in the protocol.
* Female patients must be postmenopausal (for at least one year and confirmed by serum FSH at screening), or surgically sterile, practicing true sexual abstinence, or using Investigator-approved methods of contraception throughout the study until after the post study physical examination and have a negative pregnancy test at screening.
* Sexually active male patients must use condoms with their partners throughout the study and for 90 days after completion of the study in addition to their partner's normal mode of contraception.
* Male patients must not donate sperm during the study and for 90 days after the completion of the study.
* Patients taking any continuous medication need to have been on a stable regimen for at least 1 month prior to Visit 1 - Screening Visit.

Exclusion Criteria:

* External anal sphincter disruption related to faecal incontinence caused by trauma.
* Patients with complicating gastrointestinal (GI) disease including those with inflammatory bowel diseases, patients that have received radiotherapy or surgery for anal cancer, patients with rectal prolapse, transanal surgery.
* Relevant history of or presence of any significant or uncontrolled cardiovascular risk including:

  1. Systolic > 160mmHg or Diastolic > 100mmHg. Patients on a stable regimen for > 3 months with controlled hypertension prior to Visit 1 - Screening Visit (Systolic < 140mmHg or Diastolic < 90mmHg) can be included.
  2. Abnormal 24 hour Screening Holter: corrected QT interval (QTcf) prolongation with cut-off values of >460 ms for females and >430 ms for males, acute arrhythmia, nocturnal bradycardia with heart rate (HR) < 40bpm, atrial fibrillation, AV block Type II and III, Sick Sinus Syndrome, vasovagal syncope.
  3. Fixed cardiac output states (severe aortic stenosis (AS), hypertrophic obstructive cardiomyopathy (HOCM).
  4. Significant mitral regurgitation (MR).
  5. Cardiac failure (New York Heart Association (NYHA) stage II-IV).
* Severe or uncontrolled asthma or chronic obstructive pulmonary disease determined by clinical history, physical examination, lung function tests or exercise tolerance
* Chronic liver disease (e.g. liver cirrhosis, chronic hepatitis, severe hepatic insufficiency).
* Vascular claudication after <50 metres walking distance.
* Severe renal impairment defined as glomerular filtration rate (GFR) ≤ 30 ml/min, uncontrolled and reno-vascular end stage renal disease.
* Patients with diabetic polyneuropathies.
* Any type of chronic diarrhoea or frequent diarrhoea (defined as >5 loose stools per day).
* Faecal impaction and overflow diarrhoea.
* Male patients with clinically diagnosed prostatic hyperplasia.
* Clinically significant electrolyte abnormalities, e.g. clinically significant low/high potassium and low sodium.
* Presence of clinical symptomatic haemorrhoids (grade III and IV), anal fissures or anorectal fistulas.
* Less than 2 episodes of faecal incontinence (solids, liquid, gas or mucus) per week during the 4 week historical period prior to Visit 1 - Screening Visit.
* Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
* Known history of allergy to methoxamine or any other ingredients of the Investigational Medicinal Product.
* Patients who, in the opinion of the Investigator, are unsuitable for participation in the study due to any dependencies, general medical conditions or significant illness within two weeks prior to randomisation.
* Use of any disallowed concomitant medication or other medication that the Investigator believes may affect the study including over-the-counter (OTC) products within 30 days prior to the Investigational Medicinal Product administration.
* A personal or family history of QTcf prolongation or sudden death.
* Patients taking Loperamide (2mg) >8 tablets per day for faecal incontinence either alone or in combination with codeine phosphate and/or paracetamol (8/500mg).
* Patients using any device for the treatment of faecal incontinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of NRL001 in faecal incontinence by assessing the improvement of the incontinence status after 4 weeks of treatment compared to baseline by means of the Wexner score | Up to 8 weeks

SECONDARY OUTCOMES:
To provide data on the efficacy of NRL001 in patients with faecal incontinence over an 8 week treatment period | 8 weeks
To provide preliminary data on the safety and tolerability of NRL001 (5mg, 7.5mg and 10mg) over an 8 week treatment period compared to placebo | 8 weeks
To evaluate the population pharmacokinetics and to establish any pharmacokinetic/pharmacodynamic relationship with adverse events | 8 weeks
To evaluate the dose-response relationship in order to identify the appropriate dose(s) of NRL001 for future studies | 8 weeks
To evaluate the effect of treatment according to the patient's Faecal Incontinence Quality of Life questionnaire at 4 and 8 weeks | 8 weeks
To evaluate the effect of treatment according to the Vaizey score at 4 and 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Siproudhis, MD, Principal Investigator — Hopital Pontchaillou
Locations (51):
- Czechia (8):
  - Fakultni Nemocnice BRNO, Brno
  - Gastroenterologie S R O, Hradec Králové
  - Krajska Nemocnice Liberec, Liberec
  - Fakulni Nemocnice Kralovske, Prague
  - Egk S.R.O Sanatoriu< Sv, Prague
  - GEP Clinic S.R.O, Prague
  - Fakultni Nemocnice V Motole, Prague
  - Fakultni Nemocnice Na Bulovce, Gynekologicko-Porodnicka Klinika, Prague
- France (5):
  - Chu Bordeaux - Hopital St Andre, Bordeaux
  - Chu Lyon Groupement Hospitalier Edouard Herriot, Lyon
  - Chu Nantes - Hotel Dieu - Institut Des Maladies De L'Appareil Digestif (IMAD), Nantes
  - Dr Laurent Siproudhis, Rennes
  - Chu Rouen - Hopital De Charles Nicolle, Rouen
- Germany (3):
  - Zentrum Fur Darm-Und Beckenchirurgie, Berlin
  - Martin-Luther-Krankenhaus, Berlin
  - Universitats-Frauenklink, Heidelberg
- Hungary (6):
  - PMC Pannon Medical Center, Budapest
  - Polyclinic for Outpatients, Szakrendelo Intezet, Budapest
  - University of Debrecen, Medical and Health Science Center, Debrecen
  - University of Szeged, Albert Szent-Gyorgyi Clinical Center, Faculty of Medicine, Szeged
  - Javorszky Odon Hopsital, Vac Argenti
  - Csolnoky Ferenc Veszprem, Veszprém
- Italy (6):
  - Chirurgia Gastroenterologica, Milan
  - Casa Di Cura San Pio X, Milan
  - Seconda Unita Operativa Di Chirurgia Generale, Pordenone
  - Dipartimento Emergenza Urgenza, Rome
  - Unita Operativa Complessa Gastroenteroloogia A, Rome
  - Unita Operativa Complessa Patologia Chirurgica A Indirizzo Gastroenterologico, Rome
- Poland (10):
  - Nzoz Vitamed, Bydgoszcz
  - General And Proctology Surgeon, Gdów
  - Centrum Medyczne, Wyzszej Szkoly Informatycznej, Głowno
  - Nzoz Mekmed S.C. Przychondnia Lekarska, Katowice
  - Nzoz Mikomed, Lodz
  - Osrodek Badawczo - Leczniczy Zbigniew Zegota, Ostróda
  - Endoskopia, Sopot
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - Lecznica Prosen SMO Private Medical Health Care Centre, Warsaw
  - Ars Medica SC, Wroclaw
- Spain (5):
  - Hospital Valle De Hebron, Barcelona
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital De Mataro, Mataró
  - USP, Hospital De Marbella, Málaga
  - Hospital Clinico Universtiaria Lozana Blesa, Zaragoza
- Sweden (4):
  - Pelvic Floor Centre, Malmo
  - Kirurgiska Kliniken Universitetssjukhuset, Örebro
  - Enheten For Nedre Abdominell Kirurgi, Stockholm
  - Institute of Surgical Sciences, Uppsala
- United Kingdom (4):
  - St Mark's Hospital, London
  - University College Hospital, London
  - Queens Medical Centre, Nottingham
  - Nothern General Hopsital, Sheffield